CLINICAL TRIAL: NCT06297226
Title: A Phase 2, Open-Label, Multicenter Study of Arlocabtagene Autoleucel (BMS-986393), a GPRC5D-directed CAR T Cell Therapy in Adult Participants With Relapsed or Refractory Multiple Myeloma (QUINTESSENTIAL)
Brief Title: Study of Arlocabtagene Autoleucel (BMS-986393) a GPRC5D-directed CAR T Cell Therapy in Adult Participants With Relapsed or Refractory Multiple Myeloma
Acronym: QUINTESSENTIAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA088-1000
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory Multiple Myeloma; Multiple Myeloma; BMS-986393; CAR T Cell Therapy; RRMM; Arlocabtagene Autoleucel
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arlocabtagene Autoleucel Cohort 1 (Experimental)
  Interventions: Biological: Arlocabtagene Autoleucel
- Arlocabtagene Autoleucel Cohort 2 (Experimental)
  Interventions: Biological: Arlocabtagene Autoleucel

INTERVENTIONS:
Biological: Arlocabtagene Autoleucel — Specified dose on specified days
  Other Names: CC-95266,; GPRC5D CAR T cells; BMS-986393; Arlo-cel

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Arlocabtagene Autoleucel (BMS-986393) in participants with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria

* Documented diagnosis of multiple myeloma (MM) as per International Myeloma Working Group (IMWG) criteria.
* Received at least 4 classes of MM treatment [including immunomodulatory drug (IMiD), proteasome inhibitor (PI), anti CD38 mAb, anti-BCMA therapy, and at least 3 prior lines of therapy (LOT).
* Documented disease progression during or after their last anti-myeloma regimen as per IMWG 2016 criteria.
* Participants must have measurable disease during screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria

* Active or history of central nervous system involvement with MM.
* Active systemic fungal, bacterial, viral, or other infection despite appropriate anti-infective treatment at the time of leukapheresis. Participants with severe infection, severe sepsis or bacteremia in the last 28 days prior to leukapheresis are excluded.
* Received any prior therapy directed at G protein-coupled receptor class C, group 5, member D (GPRC5D) or has received other prior treatment for MM without the required washout prior to leukapheresis.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Best overall response (BOR) of partial response (PR) or better | Up to approximately 5 years
  The number and percent of participants achieving BOR of partial response (PR) or better in quadruple class exposed participants received at least 4 prior lines of therapy (LOT)

SECONDARY OUTCOMES:
BOR of partial response (PR) or better | Up to approximately 5 years
  The number and percent of participants achieving BOR of PR in quadruple class exposed participants received at least 3 prior LOT
Best overall response (BOR) of complete response (CR) including stringent complete response (sCR) | Up to approximately 5 years
  The number and percent of participants achieving complete response (CR) [including stringent complete response sCR] in participants having received at least 3 prior lines of therapy (LOT)
Minimal residual disease (MRD) negative status | Up to approximately 5 years
Time from BMS-986393 infusion to first documentation of response of partial response (PR) or better according to the International Myeloma Working Group (IMWG) Response Criteria assessed by an independent review committee (IRC) | Up to approximately 5 years
Duration of response (DOR) assessed by an IRC | Up to approximately 5 years
  Median DOR for responders only as estimated using Kaplan-Meier method and frequencies of participants who progressed, died, and were censored
Progression-free survival (PFS) | Up to approximately 5 years
Overall survival (OS) | Up to approximately 5 years
Overall response rate (ORR) assessed by an Investigator | Up to approximately 5 years
Complete response rate (CRR) assessed by an Investigator | Up to approximately 5 years
Time to response (TTR) assessed by an Investigator | Up to approximately 5 years
Duration of response (DOR) assessed by an Investigator | Up to approximately 5 years
Progression-free survival (PFS) with BOR according to the IMWG Response Criteria assessed by Investigator | Up to approximately 5 years
Maximum observed plasma concentration (Cmax) | Up to approximately 5 years
Area under the concentration-time curve (AUC) | Up to approximately 5 years
Time of maximum observed plasma concentration (Tmax) | Up to approximately 5 years
Mean changes from baseline in European Organization for Research and Treatment of Cancer - Quality of Life C30 (EORTC QLQ-C30) selected subscales | Up to approximately 5 years
Incidence of healthcare resource utilization (HCRU) events during treatment and during post-treatment follow-up | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (52):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 214), Los Angeles, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Local Institution - 0065, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Local Institution - 0067, Charlotte, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Local Institution - 0070, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution - 0069, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Methodist HealthCare System of San Antonio Clinical Trials Office, Texas Transplant Institute, San Antonio, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - McGill University Health Centre, Montreal, Quebec
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Chiba University Hospital, Chiba
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Japanese Red Cross Medical Center, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06297226.html